CLINICAL TRIAL: NCT00001527
Title: Role of Endothelin in the Regulation of Vascular Tone in Patients With Essential Hypertension
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960016; 96-H-0016
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-11

CONDITIONS: Hypertension
Keywords: BQ-123; BQ-788; Endothelin; Endothelium; Plethysmography; Essential Hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension

SUMMARY:
Endothelin-1 (ET-1) is a powerful vasoconstricting peptide produced predominantly by vascular endothelial cells, that exerts its effect through the interaction with specific receptors, ETA and ETB, on the underlying smooth muscle cells. Previous studies in normal subjects have demonstrated an increase in forearm blood flow after ET-1 antagonism, suggesting a physiologic role of ET-1 in the regulation of basal vascular tone. However, whether ET-1-mediated tone is increased in hypertensive patients is unknown.

The main purpose of this study will be to compare the forearm vascular responses to local infusion of ET-1 receptor antagonists between normotensive and hypertensive subjects in order to assess whether ET-1-mediated basal tone is increased in patients with hypertension. In addition, we propose to study the vascular responses to local ET-1 infusion to determine whether vascular smooth muscle sensitivity to this peptide is increased in hypertensive vessels. We will use both an ETA receptor antagonist, BQ-123, and an ETB receptor antagonist, BQ-788, in order to evaluate the relative contribution of the two receptor subtypes to the regulation of vascular tone.

All drugs will be infused into the brachial artery and the responses of the forearm vasculature will be measured by means of strain gauge plethysmography. Because of the relative long-lasting effect of most of the substances to be infused, the study will be performed on two separate occasions.

DETAILED DESCRIPTION:
Endothelin-1 (ET-1) is a powerful vasoconstricting peptide produced predominantly by vascular endothelial cells, that exerts its effect through the interaction with specific receptors, ETA and ETB, on the underlying smooth muscle cells. Previous studies in normal subjects have demonstrated an increase in forearm blood flow after ET-1 antagonism, suggesting a physiologic role of ET-1 in the regulation of basal vascular tone. However, whether ET-1-mediated tone is increased in hypertensive patients is unknown.

The main purpose of this study will be to compare the forearm vascular responses to local infusion of ET-1 receptor antagonists between normotensive and hypertensive subjects in order to assess whether ET-1-mediated basal tone is increased in patients with hypertension. In addition, we propose to study the vascular responses to local ET-1 infusion to determine whether vascular smooth muscle sensitivity to this peptide is increased in hypertensive vessels. We will use both an ETA receptor antagonist, BQ-123, and an ETB receptor antagonist, BQ-788, in order to evaluate the relative contribution of the two receptor subtypes to the regulation of vascular tone.

All drugs will be infused into the brachial artery and the responses of the forearm vasculature will be measured by means of strain gauge plethysmography. Because of the relative long-lasting effect of most of the substances to be infused, the study will be performed on two separate occasions.

ELIGIBILITY:
Between 40-65 years old.

Normal Volunteers who are not taking medications. Have no medical problems. Cholesterol below 200 mg/dl. No contraceptives.

Hypertensive Patients with blood pressure greater than 145/90 off medications. Serum cholesterol less than 200 mg/dl. No other medical problems.

High cholesterol patients with cholesterol level greater than 250 mg/dl. No other medical problems.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1995-11; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Yanagisawa M, Kurihara H, Kimura S, Tomobe Y, Kobayashi M, Mitsui Y, Yazaki Y, Goto K, Masaki T. A novel potent vasoconstrictor peptide produced by vascular endothelial cells. Nature. 1988 Mar 31;332(6163):411-5. doi: 10.1038/332411a0. PMID 2451132
- [Background] Rubanyi GM, Polokoff MA. Endothelins: molecular biology, biochemistry, pharmacology, physiology, and pathophysiology. Pharmacol Rev. 1994 Sep;46(3):325-415. No abstract available. PMID 7831383
- [Background] Sakurai T, Yanagisawa M, Takuwa Y, Miyazaki H, Kimura S, Goto K, Masaki T. Cloning of a cDNA encoding a non-isopeptide-selective subtype of the endothelin receptor. Nature. 1990 Dec 20-27;348(6303):732-5. doi: 10.1038/348732a0. PMID 2175397